CLINICAL TRIAL: NCT00456911
Title: Prospective Longitudinal Study on Health and Diet (Etude Longitudinale Prospective Alimentation et Santé)
Brief Title: Family Dietary Coaching to Improve Nutritional Intakes and Body Weight Control
Acronym: ELPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Documentation du Sucre (Other)
Collaborators: Ministry of Higher Education and Research, France (Other Government); Paris Academy (Rectorat de Paris) (Unknown); Avenance Enseignement (Unknown); Fondation Louis Bonduelle (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: ELPAS 2002-RN31
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Last update posted 2008-02-13 (Estimated); Status verified 2007-04

CONDITIONS: Primary Prevention; Obesity Prevention; Body Weight Control
Keywords: obesity; prevention; children; adults; family; dietary; coaching; body mass index; fat mass
MeSH Terms: conditions — Obesity | interventions — CD36 Antigens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Fat and carbohydrate controlled diet

SUMMARY:
We hypothesize that Family Dietary Coaching for one school year will allow a nutritional shift towards following recommendations and improve health indicators in free-living children and adults.

DETAILED DESCRIPTION:
Insufficient evidence supports the feasibility and the efficacy of current nutritional recommendations to prevent obesity. The purpose of this study is to test the hypothesis that family dietary coaching would improve nutritional intakes and health indicators in free-living children and adults.

Intervention: the 1013 participating families (1013 children and 1013 parents) are randomly assigned to Group A (advice to reduce fat and to increase complex carbohydrates), Group B (advice to reduce both fat and sugars and to increase complex carbohydrates) or a control group (no advice). GA and GB receive monthly phone counseling and Internet-based monitoring. Main outcome measures are changes in nutritional intakes and body mass index throughout the intervention in both children and adults. Secondary outcomes included changes in fat mass, physical activity, fasting blood indicators and food-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* second- or third-grade pupils
* affiliation with the French Health Care System
* written informed consent

Exclusion Criteria: no inclusion criteria were based on pathological, ethnical or socio-educative indicators

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2020
Dates: Start 2005-03; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
changes in body mass index throughout the intervention

SECONDARY OUTCOMES:
changes in nutritional intakes throughout the intervention
changes in fat mass throughout the intervention
changes in anthropometric indicators throughout the intervention
changes in physical activity throughout the intervention
changes in fasting blood indicators throughout the intervention (adults only)
changes in food-related quality of life throughout the intervention (adults only)

CONTACTS AND LOCATIONS:
Overall Officials: Alain BOULIER, MD, PHD, Study Chair — Department of Nutrition and Functional Investigations, INSERM U695, Bichat-Claude Bernard Hospital, Paris, France; Dominique-Adèle CASSUTO, MD, Study Chair — Paris, France; Judith CHWALOW, PHD, Study Chair — Department of Nutrition, EA3502, Hôtel-Dieu, Paris, France; Pierre COMBRIS, PHD, Study Chair — INRA-CORELA, Ivry-sur-Seine, France; Charles COUET, MD, Study Chair — INSERM E211, Tours Hospital, Tours, France; Béatrice JOURET, MD, Study Chair — Department of Pediatrics, Children's Hospital, Toulouse, France; Monique ROMON, MD, Study Chair — Department of Nutrition, EA2694 Lille2 University, Lille, France; Chantal SIMON, MD, PhD, Study Chair — Louis Pasteur University, Medical Faculty, EA 1801, Strasbourg, France; Maïté TAUBER, MD, Study Chair — Department of Pediatrics, Children's Hospital, Toulouse, France; Paul VALENSI, MD, Principal Investigator — Department of Endocrinology, CRNH Ile-de-France, Jean Verdier Hospital, Bondy, France; Francis BORNET, MD, PHD, Study Chair — Nutri-Health, Rueil-Malmaison, France; Damien PAINEAU, MS, Study Chair — Nutri-Health, Rueil-Malmaison, France
Locations (1):
- Free-Living Participants, Paris, Île-de-France Region, France

REFERENCES:
- [Derived] Paineau DL, Beaufils F, Boulier A, Cassuto DA, Chwalow J, Combris P, Couet C, Jouret B, Lafay L, Laville M, Mahe S, Ricour C, Romon M, Simon C, Tauber M, Valensi P, Chapalain V, Zourabichvili O, Bornet F. Family dietary coaching to improve nutritional intakes and body weight control: a randomized controlled trial. Arch Pediatr Adolesc Med. 2008 Jan;162(1):34-43. doi: 10.1001/archpediatrics.2007.2. PMID 18180410
- See also: French Ministry of Research website — http://www.sante-jeunesse-sports.gouv.fr